CLINICAL TRIAL: NCT04785482
Title: Parents Post-traumatic Stress Before and After Their Infant's Second Palliative Heart Surgery: The PaTHS Descriptive Correlational Longitudinal Study
Brief Title: The PaTHS Descriptive Correlational Longitudinal Study
Acronym: PaTHS
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Melissa Elliott, Advanced Practice Registered Nurse, Children's Mercy Hospital Kansas City
Other Study IDs: STUDY00001652
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Single-ventricle; Posttraumatic Stress Disorder; Psychosocial Impairment
Keywords: remote monitoring; nursing; parents; transition
MeSH Terms: conditions — Univentricular Heart; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents of infants with single ventricle heart disease: All participants

SUMMARY:
The primary objective of this study is to measure parent's post-traumatic stress before and after their infant's second palliative heart surgery for single ventricle congenital heart disease. The investigators will use the posttraumatic stress disorder checklist for the DSM-V (PCL-5) to measure levels 2-4 weeks before and after the infant's second heart surgery. The investigators aim to describe the levels at the two-time points, compare the scores, and identify demographic information that correlates with the scores.

ELIGIBILITY:
Inclusion Criteria:

* Parent who is 18 years or older of an infant with SVCHD
* Following with CHAMP through Children's Mercy Hospital. Any person personally identifying as a parent of the child, who lives in the same household as the infant, and who will provide primary care after discharge from the hospital is eligible to participate.

Exclusion Criteria:

* Parents of an SVCHD infant who is undergoing end-of-life care, determined by the primary care team.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents of infants with single ventricle congenital heart disease participating in the Cardiac High Acuity Monitoring Program (CHAMP)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Measure the level of parental post-traumatic stress two to four weeks before their infant's second palliative heart surgery | on average at 4-6 months of age
  Measure level using the posttraumatic stress disorder checklist for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition. The scores range 0-80 with scores greater than or equal to 31 suggest provisional Posttraumatic stress disorder diagnosis.

SECONDARY OUTCOMES:
Measure the level of parental post-traumatic stress two to four weeks after discharge following their infant's second palliative heart surgery. | On average 5-6 months of age
  Measure level using the posttraumatic stress disorder checklist for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition. The scores range 0-80 with scores greater than or equal to 31 suggest provisional Posttraumatic stress disorder diagnosis.

OTHER OUTCOMES:
Examine the relationship of parental post-traumatic stress level before and after their infant's second palliative heart surgery. | through study completion, an average of 1 year
  Compare the two PCL-5 scores.
Examine what demographic variables are the mediators and moderators of the correlations. | through study completion, an average of 1 year
  Examine any correlation between selected demographics and PCL-5 scores.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Elliott, Principal Investigator — Advanced Practice Registered Nurse
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No